CLINICAL TRIAL: NCT05458167
Title: HEdia eXercise Algorithm - HEXA Study. A Randomised Controlled Crossover Pilot Study
Brief Title: HEdia eXercise Algorithm - HEXA Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hedia ApS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HEXA study
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device: Hedia Diabetes Assistant with physical activity module. (Experimental): The participants will take part in a 45-minute moderate-intensity exercise bout on a stationary ergometer bike. Participants will use the Hedia Diabetes Assistant bolus calculator with the physical activity module (intervention) during a 24-hour period starting one hour before the bout of exercise.
  Interventions: Device: Hedia Diabetes Assistant bolus calculator with a physical activity module
- Usual treatment (Active Comparator): The participants will take part in a 45-minute moderate-intensity exercise bout on a stationary ergometer bike. Participants will use their habitual diabetes management approach during a 24-hour period starting one hour before the bout of exercise (control).
  Interventions: Device: Hedia Diabetes Assistant bolus calculator with a physical activity module

INTERVENTIONS:
Device: Hedia Diabetes Assistant bolus calculator with a physical activity module — Hedia Diabetes Assistant bolus calculator with a physical activity module is a software device that calculates an insulin bolus based on blood glucose, carbohydrates and physical activity.

SUMMARY:
A randomised controlled crossover pilot study to evaluate safety and efficacy of a digital insulin bolus calculator with a physical activity module

DETAILED DESCRIPTION:
Hedia Diabetes Assistant is a software device intended to monitor blood glucose and to support in the decision making of the optimal bolus insulin dose for management of insulin-dependent diabetes by providing the user with an indicative Bolus insulin dose.

This study has been designed to investigate the safety and efficacy of a digital insulin bolus calculator with a physical activity module that provides guidance on insulin reduction to patients with type 1 diabetes mellitus prior to and after exercise, based on exercise duration and intensity compared with the patients' habitual diabetes management.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Ability to understand, speak and read Danish fluently.
* Diagnosis of type 1 diabetes mellitus for ≥12 months.
* Age between ≥18 and <60 years.
* Minimum one measurement of HbA1c between 6.0 to 8.6 % (42 to 70 mmol/mol) within the last four months. If several measurements, then it is the latest one that counts.
* Body mass index (BMI) between ≥18.5 and <30 kg/m2.
* Ability to use an Apple® (iOS version 13 and up) or Android® (Android version 8.0 and up) smartphone.
* Treated with the same pen-based insulin regimen with basal insulin (insulin glargine, degludec, or detemir) and meal time insulin (insulin aspart, lispro, glulisine) for at least the three preceding months.
* Patients who can perform 45 min. of exercise at moderate intensity on an ergometer bike (investigator assessment).
* If female participants of childbearing potential; willing to have a pregnancy test performed and to use a highly effective method of contraception.

Exclusion Criteria:

* Already using Hedia Diabetes Assistant.
* Use of human insulin or premixed insulin.
* Blood pressure > 180/105 mmHg.
* Treatment with sodium-glucose transporter 2-inhibitors, glucagon-like peptide 1 receptor agonists, or glucocorticoids.
* Job situation entailing night shifts.
* Fever.
* A mental state impeding compliance with the protocol.
* Expected non-compliance with the protocol at the discretion of the principal investigator.
* Pregnancy.
* Breast-feeding.
* Dialysis therapy or eGFR < 60 ml/min.
* Patients diagnosed with claudicatio intermittens, heart failure, ischaemic heart disease or stroke.
* Patients prescribed with beta blockers.
* Abuse of alcohol or drugs in the past two years.
* On-going participation, or participation within the last 3 months, in an organised clinical study in which participants received study medication (investigator assessment).
* Surgery scheduled for the study duration period.
* An episode of diabetic ketoacidosis or severe hypoglycaemia requiring third-party assistance within the preceding 6 months.
* Known gastroparesis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Time-in-range of Hedia Diabetes Assistant bolus calculator with physical activity module | 24-hour period starting one hour before exercise
  To compare the efficacy of the physical activity module as part of the Hedia Diabetes Assistant bolus calculator compared to the participants' habitual diabetes management during a 24-hour period starting one hour before exercise in adults with type 1 diabetes mellitus in terms of time-in-range (blood glucose 3.9-10.0 mmol/l).

SECONDARY OUTCOMES:
Hypoglycemic events of Hedia Diabetes Assistant bolus calculator with physical activity module | 24-hour period starting one hour before exercise
  To compare the efficacy of the physical activity module as part of the Hedia Diabetes Assistant bolus calculator compared to the participants' habitual diabetes management during a 24-hour period starting one hour before exercise in adults with type 1 diabetes mellitus in terms of no. of hypoglycemic events (blood glucose < 3.9 mmol/l).
Time-above-range of Hedia Diabetes Assistant bolus calculator with physical activity module | 24-hour period starting one hour before exercise
  To compare the efficacy of the physical activity module as part of the Hedia Diabetes Assistant bolus calculator compared to the participants' habitual diabetes management during a 24-hour period starting one hour before exercise in adults with type 1 diabetes mellitus in terms of time-above-range (>10.0 mmol/l).
Time-below-range of Hedia Diabetes Assistant bolus calculator with physical activity module | 24-hour period starting one hour before exercise
  To compare the efficacy of the physical activity module as part of the Hedia Diabetes Assistant bolus calculator compared to the participants' habitual diabetes management during a 24-hour period starting one hour before exercise in adults with type 1 diabetes mellitus in terms of time-below-range (blood glucose < 3.9 mmol/l).

OTHER OUTCOMES:
Glycemic variability of Hedia Diabetes Assistant bolus calculator with physical activity module | 24-hour period starting one hour before exercise
  To compare the efficacy of the physical activity module as part of the Hedia Diabetes Assistant bolus calculator compared to the participants' habitual diabetes management during a 24-hour period starting one hour before exercise in adults with type 1 diabetes mellitus in terms of glycaemic variability (coefficient of variation and standard deviation).
Daily insulin requirement of Hedia Diabetes Assistant bolus calculator with physical activity module | 24-hour period starting one hour before exercise
  To compare the daily intake of insulin in adults with type 1 diabetes mellitus utilising the physical activity module as part of the Hedia Diabetes Assistant bolus calculator compared to their habitual diabetes management during a 24-hour period starting one hour before exercise.
Daily correctional actions of Hedia Diabetes Assistant bolus calculator with physical activity module | 24-hour period starting one hour before exercise
  To compare the number of daily correctional actions (intake of food or injection of insulin) in adults with type 1 diabetes mellitus utilising the physical activity module as part of the Hedia Diabetes Assistant bolus calculator compared to their habitual diabetes management during a 24-hour period starting one hour before exercise.
Usability of Hedia Diabetes Assistant bolus calculator with physical activity module | 1 day
  To compare the usability of the physical activity module as part of the Hedia Diabetes Assistant application by System Usability Scale (SUS) in adult patients with type 1 diabetes mellitus.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Østerskov, Study Director — Hedia ApS
Locations (1):
- North Zealand Hospital - Hillerød, Hillerød, Denmark